CLINICAL TRIAL: NCT07236463
Title: Performance and Safety of Labile Iron Removal by Adding the Iron Chelator MEX-CD1 to Dialysate During Continuous Veno-venous Hemodialysis for Sepsis-associated AKI: Protocol for a Phase I-II Randomized Crossover Pilot Study.
Brief Title: Labile Iron Removal by Adding the Iron Chelator MEX-CD1 to Dialysate in Sepsis-Associated Acute Kidney Injury
Acronym: IRON-IC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIMAO/2023-1/SB-01
Record Dates: First submitted 2025-08-21; First posted 2025-11-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury; Sepsis
Keywords: Acute Kidney Injury; Sepsis; Continuous Renal Replacement Therapy; Iron Chelating Agents; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of two treatment sequences using a computer-generated, block-randomized list prepared by an independent statistician.
  * Sequence A: MEX-CD1-supplemented dialysate first, then standard dialysate
  * Sequence B: Standard dialysate first, then MEX-CD1-supplemented dialysate
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A: MEX-CD1-supplemented dialysate first, then standard dialysate (Other): Participants will receive two consecutive 24-hour CVVHD sessions using:
  * Standard Dialysate: Commercially available CiCa™ dialysate (Fresenius Medical Care, Germany)
  * MEX-CD1 Dialysate: CiCa™ dialysate supplemented with MEX-CD1 at 50 mg/L (28). MEX-CD1 remains confined to the dialysate, separated from the patient's circulation by the dialysis membrane because of its molecular weight
  Interventions: Combination Product: Continuous veino-veinous dialysis with iron-chelator supplemented dialysate
- Sequence B: Standard dialysate first, then MEX-CD1-supplemented dialysate (Other): Participants will receive two consecutive 24-hour CVVHD sessions using:
  * Standard Dialysate: Commercially available CiCa™ dialysate (Fresenius Medical Care, Germany)
  * MEX-CD1 Dialysate: CiCa™ dialysate supplemented with MEX-CD1 at 50 mg/L (28). MEX-CD1 remains confined to the dialysate, separated from the patient's circulation by the dialysis membrane because of its molecular weight
  Interventions: Combination Product: Continuous veino-veinous dialysis with iron-chelator supplemented dialysate

INTERVENTIONS:
Combination Product: Continuous veino-veinous dialysis with iron-chelator supplemented dialysate — Participants will receive two consecutive 24-hour CVVHD sessions using:
  * Standard Dialysate: Commercially available CiCa™ dialysate (Fresenius Medical Care, Germany)
  * MEX-CD1 Dialysate: CiCa™ dialysate supplemented with MEX-CD1 at 50 mg/L (28). MEX-CD1 remains confined to the dialysate, separated from the patient's circulation by the dialysis membrane because of its molecular weight
  Both sessions will use identical RRT parameters, no dose escalation is planned:
  * Continuous veno-venous hemodialysis (CVVHD) modality
  * Multifiltrate™ dialyzer (Fresenius Medical Care, Germany) with regional citrate anticoagulation
  * Dialysis dose of 20-25 mL/kg/h (approx. 1600 mL/h dialysate flow)
  * Blood flow 80 mL/min
  * Ultrasound-guided placement of a 15 cm 16 F double-lumen catheter in the right internal jugular vein
  * The circuit and the dialysis filter will be changed after each 24 hours CVVHD session

SUMMARY:
The goal of this clinical trial is to learn if adding the iron-binding drug MEX-CD1 to dialysis fluid can help remove excess iron in adults with sepsis-associated acute kidney injury (AKI) requiring dialysis who are in the intensive care unit (ICU). The main questions it aims to answer are:

Does adding MEX-CD1 to the dialysis fluid increase the amount of iron removed during dialysis? Is using MEX-CD1 in dialysis fluid safe for patients?

Participants will:

Be adults in the ICU with sepsis-associated AKI who need continuous dialysis (renal replacement therapy) Receive two 24-hour dialysis sessions: one with standard dialysis fluid and one with dialysis fluid containing MEX-CD1 Serve as their own control, meaning they will receive both treatments

Researchers will measure:

The amount of iron removed in the dialysis waste fluid (primary outcome) Blood levels of iron Changes in other trace elements Markers of inflammation and oxidative stress Safety outcomes up to 28 days after treatment This is a pilot study being done at a single hospital in France.

DETAILED DESCRIPTION:
Sepsis-associated acute kidney injury (AKI) is a common and serious complication in critically ill patients admitted to intensive care units (ICUs). It is associated with high rates of death and long-term health problems. Currently, there is no specific treatment to address the underlying causes of this condition beyond supportive measures such as dialysis to replace kidney function.

A growing body of research suggests that excess circulating labile (easily reactive) iron plays an important role in the development of organ injury during sepsis. Labile iron can promote oxidative stress, mitochondrial damage, and cell death through a process called ferroptosis. Reducing the amount of labile iron in the bloodstream may help limit these harmful effects.

This study is designed to evaluate a new approach to lowering labile iron levels during continuous renal replacement therapy (CRRT) in patients with sepsis-associated AKI. The investigational strategy uses an iron-binding compound (iron chelator) called MEX-CD1 added to the dialysis fluid (dialysate) during continuous veno-venous hemodialysis (CVVHD). By binding iron in the dialysis circuit, the chelator aims to enhance the removal of labile iron from the patient's blood without requiring systemic administration of the chelating agent.

This is a single-centre, randomised, open-label, two-period crossover phase I-II pilot study conducted in the ICU of Nîmes University Hospital in France. Each participant will undergo two consecutive 24-hour sessions of CVVHD, one using standard dialysate and one using dialysate supplemented with MEX-CD1 at a concentration of 50 mg/L. The order of the sessions will be randomised so that each participant serves as their own control, helping to reduce variability due to individual differences in illness severity or metabolism.

The primary objective of the study is to assess the performance of iron removal by measuring the concentration of iron in the dialysis effluent. Secondary objectives include evaluating plasma iron clearance, monitoring for loss of other trace elements, and assessing biomarkers related to oxidative stress and inflammation. Safety outcomes will also be closely monitored during the dialysis sessions and for 28 days afterward, including any adverse events related to the use of MEX-CD1 in the dialysate.

This pilot study will generate preliminary data on the feasibility, safety, and potential effectiveness of this novel dialysis-based iron removal strategy. If successful, it may support the development of larger trials aimed at improving outcomes for critically ill patients with sepsis-associated AKI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to ICU with sepsis-associated AKI requiring CRRT
* Sepsis defined according to SEPSIS-3 criteria (suspected/documented infection with organ dysfunction indicated by ≥2-point increase in SOFA [Sequential Organ Failure Assessment] score)
* AKI Stage 3 per KDIGO (Kidney Disease: Improving Global Outcomes) criteria: acute rise in serum creatinine ≥3 times baseline or serum creatinine ≥4 mg/dL or urine output <0.3 mL/kg/h for ≥24 hours or anuria (urine output <100ml) for ≥12 hours
* Indications for CRRT: refractory hyperkalemia (>6 mmol/L) or refractory metabolic acidosis (pH < 7.20) or acute pulmonary edema unresponsive to medical management or urine output <0.3 ml/kg/hour or anuria (urine output <100ml) persistent for 48 hours and refractory to medical treatment
* Informed consent obtained from patient or legal representative
* Affiliated with or beneficiary of a health insurance plan

Exclusion Criteria:

* Known shellfish allergy
* Moribund status with life expectancy too low to benefit
* Concurrent participation in another interventional study
* Exclusion period defined by another study
* Under legal protection (guardianship or curatorship)
* Inability to obtain informed consent from patient or representative
* Pregnant, parturient, or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Free iron concentrations in the dialysis effluent | 48 hours (2 consecutive sessions of 24 hours CVVHD)
  The primary outcome is defined as the comparison of free iron concentrations in the effluent collected during 24-hour dialysis sessions performed under two conditions: using standard dialysate and using dialysate supplemented with the iron chelator MEX-CD1.

SECONDARY OUTCOMES:
24-hour serum iron clearance | 48 hours
  24-hour serum iron clearance with iron chelation by addition of MEX-CD1 to the dialysate.
ratio iron clearance/creatinine clearance | 48 hours
  Compare the ratio of 24-hour plasma iron clearance to creatinine clearance between standard dialysate and MEX-CD1-supplemented dialysate.
Plasma malondialdehyde concentration | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on oxidative stress biomarkers by measuring plasma malondialdehyde concentrations every 8 hours for 48 hours.
Plasma Thiobarbituric Acid Reactive Substances (TBARS) | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on oxidative stress biomarkers by measuring Plasma Thiobarbituric Acid Reactive Substances (TBARS) concentrations every 8 hours for 48 hours.
Plasma protein thiols | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on oxidative stress biomarkers by measuring plasma protein thiol concentrations every 8 hours for 48 hours.
Plasma Glutathione Peroxidase (GPx) concentration | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on oxidative stress biomarkers by measuring plasma Glutathione Peroxidase (GPx) concentrations every 8 hours for 48 hours.
Plasma C-reactive protein levels | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on inflammatory biomarkers by measuring plasma C-reactive protein levels every 8 hours for 48 hours.
Plasma procalcitonin levels | From enrollment until the end of the intervention at 48 hours.
  The impact of iron chelation, achieved by adding MEX-CD1 to the dialysate, will be assessed on inflammatory biomarkers by measuring plasma procalcitonin levels every 8 hours for 48 hours.

OTHER OUTCOMES:
Number of participants with potentially treatment-related adverse events, as assessed by CTCAE v6.0, during the intervention. | From enrollment until the end of the intervention at 48 hours.
  Safety will be assessed by the incidence of potentially treatment-related adverse events during the first 48 hours of renal replacement therapy with standard dialysate or dialysate supplemented with MEX-CD1, including hypotension, cutaneous erythema, and other non-prespecified events, classified according to CTCAE v6.0.
Number of participants with potentially treatment-related adverse events, as assessed by CTCAE v6.0, after the intervention. | From the end of the intervention at Hour 48 until Day 28 or ICU discharge, whichever occurs first
  Long-term safety will be assessed by the incidence of potentially treatment-related adverse events occurring after the first 48 hours of the intervention (renal replacement therapy with standard dialysate or dialysate supplemented with MEX-CD1) and up to day 28, including anemia, low serum iron levels, and other non-prespecified events, classified according to CTCAE v6.0.
Serum iron levels | 28 Days
  the investigators will evaluate the impact of iron chelation (by adding MEX-CD1 to the dialysate) on iron balance up to Day 28. Serum iron will be measured at Day 0, Day 1, Day 2, Day 7, and Day 28."
Serum transferrin levels | 28 days
  the investigators will evaluate the impact of iron chelation (by adding MEX-CD1 to the dialysate) on iron metabolism markers up to Day 28. Serum transferrin levels will be measured at Day 0, Day 1, Day 2, Day 7, and Day 28.
Serum ferritin levels | 28 days
  the investigators will evaluate the impact of iron chelation (by adding MEX-CD1 to the dialysate) on iron metabolism markers up to Day 28. Serum ferritin levels will be measured at Day 0, Day 1, Day 2, Day 7, and Day 28.
Serum soluble transferrin receptor (sTfR) levels | 28 days
  the investigators will evaluate the impact of iron chelation (by adding MEX-CD1 to the dialysate) on iron metabolism markers up to Day 28. Serum soluble transferrin receptor (sTfR) levels will be measured at Day 0, Day 1, Day 2, Day 7, and Day 28.
Serum hepcidin levels | 28 days
  the investigators will evaluate the impact of iron chelation (by adding MEX-CD1 to the dialysate) on iron metabolism markers up to Day 28. Serum hepcidin levels will be measured at Day 0, Day 1, Day 2, Day 7, and Day 28.
24-hour copper clearance | 48 hours
  Measurement of 24-hour copper clearance after a dialysis session with MEX-CD1 added to the dialysate or with standard dialysate. Copper clearance will be calculated as: (effluent copper concentration × effluent volume over 24 hours) / serum copper concentration.
24-hour selenium clearance | 48 hours
  Measurement of 24-hour selenium clearance after a dialysis session with MEX-CD1 added to the dialysate or with standard dialysate. Selenium clearance will be calculated as: (effluent selenium concentration × effluent volume over 24 hours) / serum selenium concentration.
24-hour plasma zinc clearance | 48 hours
  Measurement of 24-hour zinc clearance after a dialysis session with MEX-CD1 added to the dialysate or with standard dialysate. Zinc clearance will be calculated as: (effluent zinc concentration × effluent volume over 24 hours) / serum zinc concentration.
24-hour aluminium clearance | 48 hours
  Measurement of 24-hour aluminium clearance after a dialysis session with MEX-CD1 added to the dialysate or with standard dialysate. Aluminium clearance will be calculated as: (effluent aluminium concentration × effluent volume over 24 hours) / serum aluminium concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Saber D BARBAR, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Nimes University Hospital, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grange C, Lux F, Brichart T, David L, Couturier A, Leaf DE, Allaouchiche B, Tillement O. Iron as an emerging therapeutic target in critically ill patients. Crit Care. 2023 Dec 4;27(1):475. doi: 10.1186/s13054-023-04759-1. PMID 38049866
- [Background] Natuzzi M, Grange C, Grea T, Brichart T, Aigle A, Bechet D, Hautefeuille B, Thomas E, Ayoub JY, Bonnet JM, Louzier V, Allaouchiche B, Couturier A, Montembault A, de Oliveira PN, David L, Lux F, Tillement O. Feasibility study and direct extraction of endogenous free metallic cations combining hemodialysis and chelating polymer. Sci Rep. 2021 Oct 7;11(1):19948. doi: 10.1038/s41598-021-99462-y. PMID 34620952
- [Derived] Couturier A, Serrand C, Masseguin C, Allaouchiche B, Tillement O, Lefrant JY, Barbar SD. Evaluation of the performance and safety of adding the iron chelator MEX-CD1 to dialysate during continuous veno-venous haemodialysis for removing excess labile iron in intensive care patients with sepsis-associated acute kidney injury - the Iron in Intensive Care trial (IRON-I.C.): protocol for a phase I-II randomised crossover pilot study. BMJ Open. 2025 Dec 23;15(12):e109783. doi: 10.1136/bmjopen-2025-109783. PMID 41436269